CLINICAL TRIAL: NCT00449878
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled Clinical Study Evaluating the Efficacy and Safety of ALTU-135 Treatment in Patients With Cystic Fibrosis-Related Exocrine Pancreatic Insufficiency
Brief Title: Liprotamase Efficacy Trial in Patients With Cystic Fibrosis-Related Exocrine Pancreatic Insufficiency
Acronym: DIGEST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anthera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14293; I5L-MC-TCAB (Other: Eli Lilly and Company); 726 (Other: Altus/Alnara)
Record Dates: First submitted 2007-03-19; First posted 2007-03-21 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Cystic Fibrosis; Exocrine Pancreatic Insufficiency
Keywords: cystic fibrosis-related pancreatic insufficiency
MeSH Terms: conditions — Cystic Fibrosis; Exocrine Pancreatic Insufficiency | interventions — liprotamase lipase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liprotamase (Experimental): Liprotamase is a fixed combination of lipase (32,500 units), protease (25,000 units) and amylase (3,750 units).
  Open Label Period: Liprotamase administered orally with each of three meals and two snacks daily for 21 days.
  Double Blind Treatment Period: Administered orally with each of three meals and two snacks daily for 6 days.
  Second Open Label Period: Administered orally with each of three meals and two snacks daily for 7 days.
  Interventions: Drug: Liprotamase
- Placebo (Placebo Comparator): Double Blind Treatment Period: Placebo (microcrystalline cellulose) administered orally with each of three meals and two snacks daily for 6 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liprotamase — Administered orally
  Other Names: ALTU-135; LY3031642; TheraCLEC - Total
  Arms: Liprotamase
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
This is a clinical trial which will evaluate the efficacy of Liprotamase treatment in cystic fibrosis (CF) patients with exocrine pancreatic insufficiency (PI).

DETAILED DESCRIPTION:
This trial is divided into four distinct periods:

1. Baseline Period during which each patient is taken off pancreatic enzyme medications.
2. An Open-Label Treatment Period during which all patients will receive ALTU-135 (liprotamase).
3. Inpatient, Double Blind Treatment Period during which half of patients will be withdrawn from treatment and will receive Placebo.
4. Second Open-Label Treatment Period during which all patients will resume treatment with ALTU-135 (liprotamase).

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential must be willing to use birth control
* Diagnosis of CF based upon the following criteria:

  * two clinical features consistent with CF; and

    * either genotype with two identifiable mutations consistent with CF, OR
    * sweat chloride >60 mEq/L by quantitative pilocarpine iontophoresis
* Clinically stable with no evidence of acute upper or lower respiratory tract infection
* PI determined by fecal elastase <100 µg/g stool measured at screening
* Able to take pancreatic enzyme supplementation in the form of capsules
* Able to perform the testing (e.g., stool collections) and inpatient stays required for this study, as judged by the Investigator
* Baseline coefficient of fat absorption (CFA) less than or equal to 80%

Exclusion Criteria:

* CFA >80% at Baseline
* Pregnancy, breastfeeding or of childbearing potential and not willing to use birth control during the study
* History of fibrosing colonopathy
* History of liver transplant, lung transplant or significant surgical resection of the bowel
* Any acute or chronic diarrheal illness unrelated to PI
* Unable to discontinue enteral tube feedings during the study
* Known hypersensitivity to food additives
* Inability to consume the diet required by the study, in the judgment of the Investigator
* Participation in an investigational study of a drug, biologic, or device not currently approved for marketing within 30 days prior to screening
* Abnormal liver function (except for patients with Gilbert Syndrome)
* Signs and/or symptoms of liver cirrhosis, portal hypertension or documented liver disease unrelated to CF
* Distal intestinal obstruction syndrome (DIOS) in the last six months prior to screening
* Unable to discontinue the use of pancreatic enzymes
* Any condition that the Investigator believes would interfere with the intent of this study or would make participation not in the best interest of the patient
* Patient is unlikely to complete the study, as determined by the Investigator

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2007-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Change from open label baseline to end of 6 day double blind treatment period in Coefficient of Fat Absorption (CFA) | Open label baseline, end of 6 day double blind treatment period

SECONDARY OUTCOMES:
Change from open label baseline to end of 6 day double blind treatment period in Coefficient of nitrogen absorption (CNA) | Open label baseline, end of 6 day double blind treatment period
Change from open label baseline to end of 6 day double blind treatment period in number of stools | Open label baseline, end of 6 day double blind treatment period
Change from open label baseline to end of 6 day double blind treatment period in stool weight | Open label baseline, end of 6 day double blind treatment period
Change from open label baseline to end of 6 day double blind treatment period in maximum blood glucose | Open label baseline, end of 6 day double blind treatment period

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stanford, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Denver, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glenview, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iowa City, Iowa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grand Rapids, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kalamazoo, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jackson, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hanover, New Hampshire
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buffalo, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cleveland, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dayton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sioux Falls, South Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Morgantown, West Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milwaukee, Wisconsin

REFERENCES:
- [Derived] Somaraju URR, Solis-Moya A. Pancreatic enzyme replacement therapy for people with cystic fibrosis. Cochrane Database Syst Rev. 2020 Aug 5;8(8):CD008227. doi: 10.1002/14651858.CD008227.pub4. PMID 32761612